CLINICAL TRIAL: NCT04536844
Title: Telehealth Follow-up in Patients With Rheumatoid Arthritis. A Noninferiority Randomized Control Trial
Brief Title: Telehealth Follow-up in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: London School of Economics and Political Science (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Anne Bull Haaversen, Co-principal Investigator, Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 33172
Record Dates: First submitted 2019-11-17; First posted 2020-09-03 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis; Treatment Compliance
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Compliance

STUDY DESIGN:
Intervention Model Description: This is a pragmatic noninferiority randomized controlled trial (RCT) in Norwegian RA patients in clinical remission (based on RAPID3 score). The patients will be allocated to 2 groups. One group will be followed up by an electronic app, while the second group will attend conventional prescheduled visits in the outpatient clinic of Martina Hansens Hospital. A computer-generated random number sequence will be used for the randomization of the RA patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth follow-up group (Experimental): Rheumatoid arthritis patients in remission who will be followed by an electronic app
  Interventions: Device: Mobile application MyDignio (follow disease activity by assigning questionnaires to participants)
- Conventional follow-up group (Placebo Comparator): Rheumatoid arthritis patients in remission who will attend conventional prescheduled visits in the outpatient clinic
  Interventions: Other: Conventional prescheduled follow-up

INTERVENTIONS:
Device: Mobile application MyDignio (follow disease activity by assigning questionnaires to participants) — An electronic application available both on Apple store and Android play which the patients can download for free will be used to collect data from the Telehealth follow up group. This group will be compared to conventional outpatient clinic follow-up group.
  Arms: Telehealth follow-up group
Other: Conventional prescheduled follow-up — Patients will be followed in the outpatient clinic by prescheduled follow-up
  Arms: Conventional follow-up group

SUMMARY:
The main objective of the present project is to test the effect of a customized Patient-Reported-Outcome (PRO)-based telehealth follow-up compared to a conventional pre-scheduled outpatient follow-up to monitor disease activity and expenses associated with the follow-up in patients with RA

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory joint disease with a high burden both for the patient and society. Outcomes for the individuals living with RA have been improved and the majority of RA patients are now in remission or low disease activity status. RA patients continue to be followed up by pre-scheduled visits, which may compromise accessibility for the sickest and thus, quality of care. The introduction of patient-initiated follow-up leads to a reduction in the use of outpatient clinic services without compromising outcomes. Self-monitoring and remote patient monitoring are facilitated by electronic innovative health tools. Among RA patients with low disease activity or remission, a Patient-Reported Outcome-based telehealth follow-up for tight control of disease activity in RA can achieve similar disease control as conventional outpatient follow-up and is likely to reduce the costs. Thus, the main objective of the present project is to test the effect of a customized PRO-based telehealth follow-up compared to a conventional prescheduled outpatient follow-up to monitor disease activity and expenses associated with the follow-up in Norwegian RA patients.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years
2. Fulfilling the European League against Rheumatism (EULAR) / American College of Rheumatology (ACR) 2010 classification criteria for RA
3. Being in remission (RAPID 3 score <=3)
4. Able to use the electronic app
5. Able to give informed consent

Exclusion Criteria:

1. <18 years
2. Severe cognitive failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients suffering a flare | 52 weeks
  comparison of the number of patients suffering a flare in each group (Flare is defined as a routine assessment of patient index data 3 (RAPID3) score >=3)

SECONDARY OUTCOMES:
Satisfaction rates | 52 weeks
  Compare satisfaction rates (as measured by Visual analog scale (VAS) satisfaction with the follow-up procedures) among the 2 patient groups
Clinical disease activity index (CDAI) | 52 weeks
  CDAI for both groups at baseline and at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diamantopoulos, MD, PhD, MPH, Principal Investigator — Martina Hansens Hospital
Locations (1):
- Martina Hansens Hospital, Sandvika, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Carmona L, Wolfe F, Vos T, Williams B, Gabriel S, Lassere M, Johns N, Buchbinder R, Woolf A, March L. The global burden of rheumatoid arthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1316-22. doi: 10.1136/annrheumdis-2013-204627. Epub 2014 Feb 18. PMID 24550173
- [Background] McBain H, Shipley M, Olaleye A, Moore S, Newman S. A patient-initiated DMARD self-monitoring service for people with rheumatoid or psoriatic arthritis on methotrexate: a randomised controlled trial. Ann Rheum Dis. 2016 Jul;75(7):1343-9. doi: 10.1136/annrheumdis-2015-207768. Epub 2015 Aug 19. PMID 26290587
- [Background] Haugeberg G, Hansen IJ, Soldal DM, Sokka T. Ten years of change in clinical disease status and treatment in rheumatoid arthritis: results based on standardized monitoring of patients in an ordinary outpatient clinic in southern Norway. Arthritis Res Ther. 2015 Aug 20;17(1):219. doi: 10.1186/s13075-015-0716-0. PMID 26290061
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] de Thurah A, Stengaard-Pedersen K, Axelsen M, Fredberg U, Schougaard LMV, Hjollund NHI, Pfeiffer-Jensen M, Laurberg TB, Tarp U, Lomborg K, Maribo T. Tele-Health Followup Strategy for Tight Control of Disease Activity in Rheumatoid Arthritis: Results of a Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Mar;70(3):353-360. doi: 10.1002/acr.23280. Epub 2018 Jan 23. PMID 28511288
- [Background] van Riel P, Alten R, Combe B, Abdulganieva D, Bousquet P, Courtenay M, Curiale C, Gomez-Centeno A, Haugeberg G, Leeb B, Puolakka K, Ravelli A, Rintelen B, Sarzi-Puttini P. Improving inflammatory arthritis management through tighter monitoring of patients and the use of innovative electronic tools. RMD Open. 2016 Nov 24;2(2):e000302. doi: 10.1136/rmdopen-2016-000302. eCollection 2016. PMID 27933206
- [Background] Pincus T, Yazici Y, Bergman M, Swearingen C, Harrington T. A proposed approach to recognise "near-remission" quantitatively without formal joint counts or laboratory tests: a patient self-report questionnaire routine assessment of patient index data (RAPID) score as a guide to a "continuous quality improvement" s. Clin Exp Rheumatol. 2006 Nov-Dec;24(6 Suppl 43):S-60-5; quiz S-66-73. PMID 17083765

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT04536844/Prot_SAP_000.pdf